CLINICAL TRIAL: NCT05183932
Title: Comparing the Effectiveness of Surgery Versus Stereotactic Body Radiation Therapy for Stage I Non-Small Cell Lung Cancer (SORT)
Brief Title: Surgery Versus Stereotactic Body Radiation Therapy for Stage I Non-Small Cell Lung Cancer
Acronym: SORT
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202112102; R01CA258681 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: * Participants will have standard of care lobectomy/segmentectomy/wedge resection. Decision for treatment will be made at the discretion of the treating physician.
  * PROMIS instruments include 8 domains and will be completed prior to treatment, 1 month post-treatment, 6 months post-treatment, 12 months post-treatment, 24 months post-treatment, and 36 months post-treatment
    * Bank 2.0 - Physical Function
    * Bank v1.1 - Pain Interference
    * Bank v1.0 - Fatigue
    * Bank v1.0 - Depression
    * Bank v1.0 - Anxiety
    * Bank v1.0 - Dyspnea Severity
    * Bank v2.0 - Ability to Participate in Social Roles and Activities
    * Bank v2.0 - Cognitive Function
- Stereotactic body radiotherapy (SBRT): * Participants will have standard of care 1-10 fractions of radiation therapy. Decision for treatment will be made at the discretion of the treating physician.
  * PROMIS instruments include 8 domains and will be completed prior to treatment, 1 month post-treatment, 6 months post-treatment, 12 months post-treatment, 24 months post-treatment, and 36 months post-treatment
    * Bank v2.0 - Physical Function
    * Bank v1.1 - Pain Interference
    * Bank v1.0 - Fatigue
    * Bank v1.0 - Depression
    * Bank v1.0 - Anxiety
    * Bank v1.0 - Dyspnea Severity
    * Bank v2.0 - Ability to Participate in Social Roles and Activities
    * Bank v2.0 - Cognitive Function

SUMMARY:
The development of stereotactic body radiation therapy (SBRT) for the treatment of stage I non-small cell lung cancer (NSCLC) has inspired a close partnership between thoracic surgery and radiation oncology. In this study, patients with stage I NSCLC will be screened prior to treatment and will be consented after their treatment plan has been determined. Prospectively collected patient-reported outcomes (PROs) will be collected for 3 years or for the duration of the study (whichever is shorter), as will outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I NSCLC (T1 or T2a, N0, M0) by CT performed within 90 days of screening.

  * PET/CT is required within 90 days of screening except under circumstances where the clinical picture suggests, or biopsy confirms, a low-grade adenocarcinoma.
  * Biopsy is strongly encouraged. In the event biopsy is not performed, rationale must be provided for performing empiric treatment.
  * Patients with hilar or mediastinal lymph nodes ≤ 1 cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Pre-treatment mediastinal lymph node sampling by any technique is allowed but not required. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but nondiagnostic uptake) are be eligible only if directed tissue biopsies of all abnormally identified areas are negative for cancer.
* First primary NSCLC on the ipsilateral side.
* At least 18 years of age.
* Clinically eligible for either treatment (surgical resection or SBRT). Because this is a pragmatic study and treatment decisions are at the discretion of the treating physicians and their patients, patients must be eligible for either treatment. To be considered eligible for either treatment, patients must have:

  * ECOG performance status ≤ 2
  * No home oxygen use
  * FEV1 and DLCO ≥ 40% predicted
  * No symptomatic congestive heart failure as documented by NYHA I-II functional classification
  * Been deemed operable by a thoracic surgeon, per clinical visit or review of the medical record and as documented by e-mail, tumor board, study meetings, or other acceptable source documentation. In addition to operability, the surgeon must define what anticipated surgical approach and procedure would be undertaken.
  * Been deemed treatable by a radiation oncologist with 10 or fewer fractions of SBRT, per clinical visit or review of the medical record and as documented by e-mail, tumor board, study meetings, or other acceptable source documentation. In addition to suitability for SBRT, the radiation oncologist must define which dose and fractionation would be undertaken.
* Ability to understand and willingness to sign an IRB-approved written informed consent document.
* Agrees to receive treatment for clinical stage I NSCLC (either surgical resection or SBRT).

Exclusion Criteria:

* Prior or concurrent malignancies, unless the natural history of the prior or concurrent malignancy does not have the potential to interfere with the interpretation of the results of the study.
* Clinically diagnosed or biopsy proven low-grade neuroendocrine carcinoma (carcinoid).
* Prior thoracic radiation therapy that would overlap with the lung cancer being treated on study.
* Previous chemotherapy, radiotherapy, or surgical resection specifically for the lung cancer being treated on study.
* Prior lung resection on the ipsilateral side positive for malignancy.
* Patients with central tumors requiring a sleeve lobectomy or pneumonectomy.
* "Ultra-central" lesions (defined as a lesion that directly contacts or overlaps the trachea, main bronchus, esophagus, or pulmonary vessels).
* Concurrent enrollment in a therapeutic trial for the index cancer.
* Synchronous primary lung cancer.
* Uncontrolled or symptomatic psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who meet the eligibility criteria from any of the participating sites listed.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Through 36 months post-treatment (estimated to be 36 months and 1 week)
  DFS is defined as time from the date of treatment to date of disease recurrence or death, whichever occurs earlier.
Change in patient-reported outcomes as measured by the PROMIS Bank survey | From baseline through 36 months post-treatment (estimated to be 36 months and 1 week)
  * Surveys will occur at baseline, 1 month post-treatment, 6 months post-treatment, 12 months post-treatment, 24 months post-treatment, and 36 months post-treatment
  * The PROMIS scores will be compared across the 8 pre-specified domains:
    * Cancer Bank v1.1 - Physical Function
    * Cancer Bank v1.1 - Pain Interference
    * Cancer Bank v1.0 - Fatigue
    * Cancer Bank v1.0 - Depression
    * Cancer Bank v1.0 - Anxiety
    * Bank v1.0 - Dyspnea Severity
    * Bank v2.0 - Ability to Participate in Social Roles and Activities
    * Bank v2.0 - Cognitive Function
  * PROMIS is scored 1-100 and normalizes to the population mean of 50 with each 10 being a standard deviation. A higher score indicates a worse patient-reported outcome.

SECONDARY OUTCOMES:
Cancer-specific survival (CSS) | Through 36 months post-treatment (estimated to be 36 months and 1 week)
  Cancer-specific survival (CSS) is defined as time from the date of treatment to date of cancer-related death. The alive patients without any signs or symptoms of that cancer are censored at the last follow-up.
Overall survival (OS) | Through 36 months post-treatment (estimated to be 36 months and 1 week)
  Overall survival (OS) is defined as time from the date of treatment to date of death. The alive patients are censored at the last follow-up.
Treated-related mortality | At 30 days (estimated to be 1 month and 1 week)
Number of post-treatment events (grade 3 and above) | Through 36 months post-treatment (estimated to be 36 months and 1 week)
  Post-treatment grade 3-5 events measured via CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Kozower, M.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (8):
- United States (7):
  - Emory University, Atlanta, Georgia
  - Carle Cancer Institute, Urbana, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu